CLINICAL TRIAL: NCT00856531
Title: Impairments of Oral Language in Subjects With the Möbius Sequence
Brief Title: Impairments of Oral Language in Mobius Syndrome
Acronym: Mobius
Status: Completed | Type: Observational
Sponsor: Fortaleza University (Other)
Responsible Party: Renata Cavalcante Barbosa Haguette, Hospital Infantil Albert Sabin
Other Study IDs: mobius syndrome
Record Dates: First submitted 2009-03-04; First posted 2009-03-05 (Estimated); Last update posted 2009-03-05 (Estimated); Status verified 2009-03

CONDITIONS: Möbius Sequence
Keywords: Möbius syndrome; Language; Speech, Language and Hearing Sciences
MeSH Terms: conditions — Mobius Syndrome; Language; Speech

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (15):
- 1
- 2
- 3
- 4
- 5
- 6
- 7
- 8
- 9
- 10
- 11
- 12
- 13
- 14
- 15

SUMMARY:
The Möbius syndrome constitutes a congenital disorder classically caused by genetic and environmental factors. The clinical manifestations include lesion of the facial and abducens nerves associated with limb malformations specially club foot. The speech-language manifestations include compromise of oral and deglutition, speech and language functions, secondary to cranial nerves lesions and mental retardation. The language compromise in this disorder is still not well known. In this way, the main objective of this study is to characterize the oral language in a population of fifteen subjects with Möbius syndrome with age ranging from two to thirteen years old, from both sexes, seen in one of the three main center for genetic diagnosis in the state of Ceará. The present work is a descriptive study of a cross-sectional design conducted from February to December/2002, using a clinical evaluation of language components including morphology, syntax, semantics and pragmatics. The investigators identified exclusive speech involvement in 20,0% of the subjects, language disturbance in 46,7%, speech and language disturbance in 13,3% and oral language involvement in 26,7%. The investigators conclude that the language disturbance in the Möbius syndrome presents with a variable compromise of all oral language components. The delay in linguistical development, incomprehensive speech and the deficit of constructions of sentences and narrations are constant.

DETAILED DESCRIPTION:
In this way, the main objective of this study is to characterize the oral language in a population of fifteen subjects with Möbius syndrome with age ranging from two to thirteen years old, from both sexes, seen in one of the three main center for genetic diagnosis in the state of Ceará. The present work is a descriptive study of a cross-sectional design conducted from February to December/2002, using a clinical evaluation of language components including morphology, syntax, semantics and pragmatics.

ELIGIBILITY:
Inclusion Criteria:

* Möbius syndrome
* Age ranging from two to thirteen years old.

Exclusion Criteria:

* Others diseases with impact in oral language.

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: fifteen subjects with Möbius syndrome with age ranging from two to thirteen years old, from both sexes, seen in one of the three main center for genetic diagnosis in the state of Ceará, Brazil.
Sampling Method: Non-Probability Sample
Dates: Start 2002-01; Primary Completion 2003-01 (Actual); Study Completion 2003-01 (Actual)